CLINICAL TRIAL: NCT03457727
Title: A Two Part, Randomized, Open-label, Cross Over Study in Healthy Elderly Participants to Evaluate the Relative Bioavailability of Hydrobromide Salt Tablet Formulations of Danirixin in the Fed and Fasted States, and to Evaluate the Effect of Food and Gastric Acid Secretion Suppression on Danirixin Pharmacokinetics Following Administration of Hydrobromide Salt Tablets
Brief Title: GSK1325756 Relative Bioavailability Study in Healthy Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 207573
Record Dates: First submitted 2018-03-01; First posted 2018-03-07 (Actual); Results first posted 2019-08-28 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Danirixin; Healthy; Food effect; Relative Bioavailability; Hydrobromide Salt
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — danirixin; Omeprazole

STUDY DESIGN:
Intervention Model Description: Subjects will receive danirixin reference and test formulations in a cross-over manner.
Masking Description: This will be an open-label study and blinding will not be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Subjects receiving danirixin: Part A (Experimental): Subjects will receive a single oral dose of 50 mg danirixin reference and test formulations with food and 240 mL of water in a cross-over manner.
  Interventions: Drug: Danirixin
- Subjects receiving danirixin without omeprazole: Part B (Experimental): Subjects will receive a single oral dose of 50 mg danirixin formulation (selected in Part A) in fasted or fed state in a cross-over manner.
  Interventions: Drug: Danirixin
- Subjects receiving danirixin with omeprazole: Part B (Experimental): Subjects will receive a single oral dose of 50 mg danirixin formulation (selected in Part A) along with once daily 40 mg OMP capsule in fasted or fed state in a cross-over manner.
  Interventions: Drug: Danirixin; Drug: Omeprazole

INTERVENTIONS:
Drug: Danirixin — Danirixin is being developed as a potential anti-inflammatory agent for the treatment of chronic obstructive pulmonary disorder (COPD) and other inflammatory diseases and influenza. Danirixin reference (600 mg) or test formulation (475 or 600 mg or 600 mg with 5 percent HPMC) immediate release tablets will be administered by oral route in a cross-over manner.
Drug: Omeprazole — Omeprazole is used as an antacid. OMP 40 mg delayed-release capsule will be administered by oral route to randomized subjects.
  Arms: Subjects receiving danirixin with omeprazole: Part B

SUMMARY:
This 2-part study will be carried out on healthy elderly subjects to evaluate relative bioavailability of danirixin formulations. Part A will support the selection of the formulation and Part B will assess food effect, bioavailability and pharmacokinetic (PK) profile of selected formulation from Part A. Danirixin is currently administered with food, therefore the investigation of food effect for the selected formulation could potentially enable dosing without food. Approximately 16 subjects will be included in Part A and approximately 24 subjects will be included in Part B. Both parts will include a screening phase, treatment phase with in-between washout period and a follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 65 to 80 years of age inclusive, at the Screening Visit.
* Subjects who are healthy, as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring or a subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included if the investigator and the GlaxoSmithKline (GSK) Medical Monitor agree that the finding is unlikely to introduce risk factors and will not interfere with the study procedures and objectives. Additionally, laboratory assessments that are specifically listed in the inclusion or exclusion criteria and are outside of the reference range can be repeated once during the screening period.
* Body weight >=50 kilograms (kg) and body mass index (BMI) within the range 19 - 34 kg per meter square (kg/m^2) (inclusive).
* Male or female subjects will be included. A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: Not a woman of childbearing potential (WOCBP) or a WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 60 hours after the last dose of study treatment.
* Capable of giving signed informed consent.
* AST, ALT, alkaline phosphatase and bilirubin <= 1.5 × upper limit of normal (ULN) (isolated bilirubin > 1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35 percent).
* Resting BP of <= 160/90 millimeters of mercury (mmHg), irrespective of anti-hypertensive medication status for the subject.
* Able to consume the Food and Drug Administration (FDA) defined high fat meal within 30 minutes in each of the four treatment periods where study treatment is administered in a fed state.

Exclusion Criteria:

* Significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data.
* Evidence of active or latent tuberculosis (TB) as documented by medical history and examination, chest x-rays (posterior anterior and lateral), and TB testing: either a positive tuberculin skin test [TST; defined as a skin induration <5 millimeter (mm) at 48 to 72 hours, regardless of Bacillus Calmette-Guerin (BCG) or other vaccination history] or a positive (not indeterminate) QuantiFERON®-TB Gold test.
* Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Breast cancer within the past 10 years.
* ALT >1.5x ULN
* Bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Corrected QT interval (QTc) >450 milliseconds (msec).
* Use of prescription or non-prescription drugs, including proton pump inhibitors, histamine receptor 2 antagonists, systemic antacid medications (unless these can be held during the study), vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study treatment until completion of the last study assessment , unless in the opinion of the investigator and GSK Medical Monitor, the medication will not interfere with the study procedures or compromise subject safety. Some examples of exceptions (permitted medications) are: Stable dose of anti-hypertensive medication for at least 3 months prior to the screening visit; Stable dose of lipid-lowering medications (statins or fibrates) for at least 3 months prior to the screening visit; Antacids up to 24 hours prior to dosing.
* Participation in the study would result in loss of blood or blood products in excess of 500 milliliter (mL) within 3 months.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 3 months, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Participation in a previous clinical trial with danirixin within 1 year prior to the first dosing day in the current study.
* Female Subjects: Positive urine beta-human chorionic gonadotropin (beta-hCG) test at screening.
* Presence of Hepatitis B surface antigen (HBsAg) at screening Positive Hepatitis C antibody test result at screening.
* Positive Hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study treatment.
* For potent immunosuppressive agents, presence of the Hepatitis B core antibody (HBcAb) should also lead to exclusion from the study even if HBsAg is negative.
* Positive pre-study drug/alcohol screen.
* Positive human immunodeficiency virus (HIV) antibody test.
* Regular use of known drugs of abuse.
* Regular alcohol consumption within 6 months prior to the study defined as: an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 grams of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Consumption of red wine, Seville oranges, grapefruit or grapefruit juice and/or pummelos, citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study treatment until collection of the final blood sample.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 90 days prior to screening.
* Sensitivity to heparin or heparin-induced thrombocytopenia.
* Sensitivity to any of the study treatments, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2018-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20808

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This two-part study assessed the relative bioavailability of Danirixin (DNX) tablet formulations along with effect of food and gastric acid secretion suppression on DNX pharmacokinetics. This study was conducted at a single center in the United States from 07-Mar-2018 to 25-Jul-2018.
Pre-assignment Details: Danirixin hemihydrate salt tablet formulation manufactured using roller compaction (RC) was compared to test formulations manufactured by direct compression (DC) with an excipient hydroxypropyl methylcellulose (HPMC) to evaluate the most appropriate formulation/dosing regimen. A total of 40 participants were enrolled in the study.
Groups:
- DNX 50 mg 600RC/475DC/600DC/600DC-5% HPMC in Fed State: Participants received a sequence of the following: single oral dose of 50 milligrams (mg) DNX hydrobromide (HBr) hemihydrate tablet formulation (600 mg tablet manufactured by RC [600 RC]) on Day 1 of treatment period 1, a single oral dose of 50 mg DNX HBr hemihydrate tablet formulation (475 mg tablet manufactured by DC [475 DC]) on Day 1 of treatment period 2, a single oral dose of 50 mg DNX HBr hemihydrate tablet formulation (600 DC) on Day 1 of treatment period 3 and 50 mg DNX HBr hemihydrate 600 DC tablet formulation with containing 5 percent HPMC on Day 1 of treatment period 4. All the formulations were administered in fed state (with a high fat meal). The treatment periods were separated by a washout period of 5 days.
- DNX 50mg 600RC/475DC/600DC/600DC-5% HPMC in Fasted State: Participants received a sequence of the following: single oral dose of 50 mg DNX HBr hemihydrate 600 RC on Day 1 of treatment period 1, a single oral dose of 50 mg DNX HBr hemihydrate 475 DC on Day 1 of treatment period 2, a single oral dose 50 mg DNX HBr hemihydrate 600 DC on Day 1 of treatment period 3 and a single oral dose of 50 mg DNX HBr hemihydrate 600 DC with 5 percent HPMC on Day 1 of treatment period 4. All the formulations were administered in fasted state. The treatment periods were separated by a washout period of 5 days.
- DNX 50 mg 475 DC Under Fasted/Normal/Fat Meal/ Mono-fat Meal: Participants received a sequence of the following: single oral dose of 50 mg DNX HBr hemihydrate 475 DC tablet formulation in fasted state on Day 1 of treatment period 1, a single oral dose of 50 mg DNX HBr hemihydrate 475 DC along with normal meal on Day 1 of treatment period 2, a single oral dose of 50 mg DNX HBr hemihydrate 475 DC along with high fat meal in treatment period 3, followed by a single oral dose of 50 mg DNX HBr monohydrate 475 DC with high fat meal in treatment period 4. The treatment periods were separated by a washout period of 5 days.
- DNX 50 mg 475 DC+OMP 40mg Under Fasted/Normal/Fat Meal State: Participants received a sequence of the following: single oral dose of 50 mg DNX HBr hemihydrate 475 DC in fasted state along with 40 mg omeprazole (OMP) during treatment period 1, a single oral dose of 50 mg DNX HBr hemihydrate 475 DC and 40 mg OMP along with normal meal in treatment period 2 and a single oral dose of 50 mg DNX HBr hemihydrate 475 DC and 40 mg OMP along with high fat meal in treatment period 3. The treatment periods were separated by a washout period of 5 days. OMP was administered from Day -4 of each treatment period through washout periods.
Period: Part 1, Period 1 (1 Day)
Arm/Group | DNX 50 mg 600RC/475DC/600DC/600DC-5% HPMC in Fed State | DNX 50mg 600RC/475DC/600DC/600DC-5% HPMC in Fasted State | DNX 50 mg 475 DC Under Fasted/Normal/Fat Meal/ Mono-fat Meal | DNX 50 mg 475 DC+OMP 40mg Under Fasted/Normal/Fat Meal State
Started | 8 | 8 | 0 | 0
Completed | 8 | 8 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 1, Washout Period 1 (5 Days)
Arm/Group | DNX 50 mg 600RC/475DC/600DC/600DC-5% HPMC in Fed State | DNX 50mg 600RC/475DC/600DC/600DC-5% HPMC in Fasted State | DNX 50 mg 475 DC Under Fasted/Normal/Fat Meal/ Mono-fat Meal | DNX 50 mg 475 DC+OMP 40mg Under Fasted/Normal/Fat Meal State
Started | 8 | 8 | 0 | 0
Completed | 8 | 8 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 1, Period 2 (1 Day)
Arm/Group | DNX 50 mg 600RC/475DC/600DC/600DC-5% HPMC in Fed State | DNX 50mg 600RC/475DC/600DC/600DC-5% HPMC in Fasted State | DNX 50 mg 475 DC Under Fasted/Normal/Fat Meal/ Mono-fat Meal | DNX 50 mg 475 DC+OMP 40mg Under Fasted/Normal/Fat Meal State
Started | 8 | 8 | 0 | 0
Completed | 8 | 8 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 1, Washout Period 2 (5 Days)
Arm/Group | DNX 50 mg 600RC/475DC/600DC/600DC-5% HPMC in Fed State | DNX 50mg 600RC/475DC/600DC/600DC-5% HPMC in Fasted State | DNX 50 mg 475 DC Under Fasted/Normal/Fat Meal/ Mono-fat Meal | DNX 50 mg 475 DC+OMP 40mg Under Fasted/Normal/Fat Meal State
Started | 8 | 8 | 0 | 0
Completed | 8 | 8 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 1, Period 3 (1 Day)
Arm/Group | DNX 50 mg 600RC/475DC/600DC/600DC-5% HPMC in Fed State | DNX 50mg 600RC/475DC/600DC/600DC-5% HPMC in Fasted State | DNX 50 mg 475 DC Under Fasted/Normal/Fat Meal/ Mono-fat Meal | DNX 50 mg 475 DC+OMP 40mg Under Fasted/Normal/Fat Meal State
Started | 8 | 8 | 0 | 0
Completed | 8 | 8 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 1, Washout Period 3 (5 Days)
Arm/Group | DNX 50 mg 600RC/475DC/600DC/600DC-5% HPMC in Fed State | DNX 50mg 600RC/475DC/600DC/600DC-5% HPMC in Fasted State | DNX 50 mg 475 DC Under Fasted/Normal/Fat Meal/ Mono-fat Meal | DNX 50 mg 475 DC+OMP 40mg Under Fasted/Normal/Fat Meal State
Started | 8 | 8 | 0 | 0
Completed | 8 | 8 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 1, Period 4 (1 Day)
Arm/Group | DNX 50 mg 600RC/475DC/600DC/600DC-5% HPMC in Fed State | DNX 50mg 600RC/475DC/600DC/600DC-5% HPMC in Fasted State | DNX 50 mg 475 DC Under Fasted/Normal/Fat Meal/ Mono-fat Meal | DNX 50 mg 475 DC+OMP 40mg Under Fasted/Normal/Fat Meal State
Started | 8 | 8 | 0 | 0
Completed | 8 | 8 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 2, Period 1 (1 Day)
Arm/Group | DNX 50 mg 600RC/475DC/600DC/600DC-5% HPMC in Fed State | DNX 50mg 600RC/475DC/600DC/600DC-5% HPMC in Fasted State | DNX 50 mg 475 DC Under Fasted/Normal/Fat Meal/ Mono-fat Meal | DNX 50 mg 475 DC+OMP 40mg Under Fasted/Normal/Fat Meal State
Started | 0 | 0 | 12 | 12
Completed | 0 | 0 | 12 | 12
Not Completed | 0 | 0 | 0 | 0
Period: Part 2, Washout Period 1 (5 Days)
Arm/Group | DNX 50 mg 600RC/475DC/600DC/600DC-5% HPMC in Fed State | DNX 50mg 600RC/475DC/600DC/600DC-5% HPMC in Fasted State | DNX 50 mg 475 DC Under Fasted/Normal/Fat Meal/ Mono-fat Meal | DNX 50 mg 475 DC+OMP 40mg Under Fasted/Normal/Fat Meal State
Started | 0 | 0 | 12 | 12
Completed | 0 | 0 | 12 | 11
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Period: Part 2, Period 2 (1 Day)
Arm/Group | DNX 50 mg 600RC/475DC/600DC/600DC-5% HPMC in Fed State | DNX 50mg 600RC/475DC/600DC/600DC-5% HPMC in Fasted State | DNX 50 mg 475 DC Under Fasted/Normal/Fat Meal/ Mono-fat Meal | DNX 50 mg 475 DC+OMP 40mg Under Fasted/Normal/Fat Meal State
Started | 0 | 0 | 12 | 11
Completed | 0 | 0 | 12 | 11
Not Completed | 0 | 0 | 0 | 0
Period: Part 2, Washout Period 2 (5 Days)
Arm/Group | DNX 50 mg 600RC/475DC/600DC/600DC-5% HPMC in Fed State | DNX 50mg 600RC/475DC/600DC/600DC-5% HPMC in Fasted State | DNX 50 mg 475 DC Under Fasted/Normal/Fat Meal/ Mono-fat Meal | DNX 50 mg 475 DC+OMP 40mg Under Fasted/Normal/Fat Meal State
Started | 0 | 0 | 12 | 11
Completed | 0 | 0 | 12 | 11
Not Completed | 0 | 0 | 0 | 0
Period: Part 2, Period 3 (1 Day)
Arm/Group | DNX 50 mg 600RC/475DC/600DC/600DC-5% HPMC in Fed State | DNX 50mg 600RC/475DC/600DC/600DC-5% HPMC in Fasted State | DNX 50 mg 475 DC Under Fasted/Normal/Fat Meal/ Mono-fat Meal | DNX 50 mg 475 DC+OMP 40mg Under Fasted/Normal/Fat Meal State
Started | 0 | 0 | 12 | 11
Completed | 0 | 0 | 12 | 11
Not Completed | 0 | 0 | 0 | 0
Period: Part 2, Washout Period 3 (5 Days)
Arm/Group | DNX 50 mg 600RC/475DC/600DC/600DC-5% HPMC in Fed State | DNX 50mg 600RC/475DC/600DC/600DC-5% HPMC in Fasted State | DNX 50 mg 475 DC Under Fasted/Normal/Fat Meal/ Mono-fat Meal | DNX 50 mg 475 DC+OMP 40mg Under Fasted/Normal/Fat Meal State
Started | 0 | 0 | 12 | 11
Completed | 0 | 0 | 12 | 11
Not Completed | 0 | 0 | 0 | 0
Period: Part 2, Period 4 (1 Day)
Arm/Group | DNX 50 mg 600RC/475DC/600DC/600DC-5% HPMC in Fed State | DNX 50mg 600RC/475DC/600DC/600DC-5% HPMC in Fasted State | DNX 50 mg 475 DC Under Fasted/Normal/Fat Meal/ Mono-fat Meal | DNX 50 mg 475 DC+OMP 40mg Under Fasted/Normal/Fat Meal State
Started | 0 | 0 | 12 | 0
Completed | 0 | 0 | 12 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DNX 50 mg 600RC/475DC/600DC/600DC-5% HPMC in Fed State | DNX 50mg 600RC/475DC/600DC/600DC-5% HPMC in Fasted State | DNX 50 mg 475 DC Under Fasted/Normal/Fat Meal/ Mono-fat Meal | DNX 50 mg 475 DC+OMP 40mg Under Fasted/Normal/Fat Meal State | Total
Number analyzed (Participants) | 8 | 8 | 12 | 12 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.4 (3.54) | 70.9 (4.58) | 71.3 (4.14) | 69.4 (2.68) | 70.3 (3.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 4 | 8 | 22
  Male | 4 | 2 | 8 | 4 | 18
Race/Ethnicity, Customized [Number; unit: Count of Participants]
  Black or African American | 1 | 0 | 0 | 2 | 3
  White | 7 | 8 | 12 | 10 | 37

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to Infinity (AUC [0-inf]) of Danirixin for Part 1
Description: Blood samples were collected at the indicated time points after administration of study treatment to investigate the pharmacokinetic (PK) profile of Danirixin. PK parameters were calculated by standard non-compartmental analysis using WinNonlin based on actual sampling times.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours in Part 1
Population: PK Population includes all participants for whom a PK sample was obtained and analyzed. Only those participants with data available at specified time frame were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Groups:
- 600RC High Fat: Participants received a single oral dose of DNX 50 mg HBr hemihydrate 600 RC tablet formulation along with a high fat meal
- 475DC High Fat: Participants received a single oral dose of DNX 50 mg HBr hemihydrate 475 DC tablet formulation along with high fat meal
- 600DC High Fat: Participants received a single oral dose of DNX 50 mg HBr hemihydrate 600 DC tablet formulation along with high fat meal
- 600DC 5%HPMC High Fat: Participants received a single oral dose of DNX 50 mg HBr hemihydrate 600 DC tablet with 5 percent HPMC formulation along with high fat meal
- 600RC Fasted: Participants received a single oral dose of DNX 50 mg HBr hemihydrate 600 RC tablet formulation under fasted condition
- 475DC Fasted: Participants received a single oral dose of DNX 50 mg HBr hemihydrate 475 DC tablet formulation under fasted condition
- 600DC Fasted: Participants received a single oral dose of DNX 50 mg HBr hemihydrate 600 DC tablet formulation under fasted condition
- 600DC 5%HPMC Fasted: Participants received a single oral dose of DNX 50 mg HBr hemihydrate 600 DC tablet with 5 percent HPMC formulation under fasted condition
Arm/Group | 600RC High Fat | 475DC High Fat | 600DC High Fat | 600DC 5%HPMC High Fat | 600RC Fasted | 475DC Fasted | 600DC Fasted | 600DC 5%HPMC Fasted
Number analyzed (Participants) | 5 | 7 | 7 | 6 | 6 | 7 | 8 | 8
Hours*nanograms per milliliter | 6166.7 (19.20) | 6052.9 (14.18) | 5816.4 (22.99) | 5996.1 (26.31) | 11394.6 (30.07) | 11285.7 (32.72) | 10957.4 (31.55) | 11230.8 (28.21)

2. Primary Outcome: Maximum Observed Concentration (Cmax) of Danirixin for Part 1
Description: Blood samples were collected at the indicated time points after administration of study treatment to investigate the PK profile of Danirixin. PK parameters were calculated by standard non-compartmental analysis using WinNonlin based on actual sampling times.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours in Part 1
Population: PK population. Only those participants with data available at specified time frame were analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms/milliliter
Arm/Group | 600RC High Fat | 475DC High Fat | 600DC High Fat | 600DC 5%HPMC High Fat | 600RC Fasted | 475DC Fasted | 600DC Fasted | 600DC 5%HPMC Fasted
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 7 | 8 | 8 | 8
Nanograms/milliliter | 761.5 (27.22) | 712.8 (20.53) | 762.3 (37.23) | 659.2 (47.40) | 2708.2 (26.22) | 2418.5 (27.78) | 2607.1 (30.24) | 2511.8 (24.19)

3. Primary Outcome: Number of Participants With Any Adverse Event (AE) and Serious Adverse Events (SAEs) in Part 1
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant.
Time Frame: Up to 29 days in Part 1
Population: Modified Intent-to-treat (mITT) Population includes all randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | 600RC High Fat | 475DC High Fat | 600DC High Fat | 600DC 5%HPMC High Fat | 600RC Fasted | 475DC Fasted | 600DC Fasted | 600DC 5%HPMC Fasted
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
Participants
  Any AE | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 1
  Any SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Vital Signs of Potential Clinical Concern in Part 1
Description: Vital signs included systolic and diastolic blood pressure, temperature, respiratory rate and pulse rate were measured with participants in semi-supine position after 5 minutes rest.
Time Frame: Up to 29 days in Part 1
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | 600RC High Fat | 475DC High Fat | 600DC High Fat | 600DC 5%HPMC High Fat | 600RC Fasted | 475DC Fasted | 600DC Fasted | 600DC 5%HPMC Fasted
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
Participants | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With 12-lead Electrocardiogram (ECG) Values of Potential Clinical Concern in Part 1
Description: Single 12-lead ECGs were obtained using an ECG machine that automatically calculated the heart rate and measured PR, QRS, and QT intervals, and QT interval corrected by Fridericia's formula (QTcF). Number of participants with 12-lead ECG values of potential clinical concern in Part 1 are presented.
Time Frame: Up to 29 days in Part 1
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | 600RC High Fat | 475DC High Fat | 600DC High Fat | 600DC 5%HPMC High Fat | 600RC Fasted | 475DC Fasted | 600DC Fasted | 600DC 5%HPMC Fasted
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
Participants | 1 | 2 | 2 | 2 | 2 | 1 | 2 | 1

6. Primary Outcome: Number of Participants With Laboratory Values of Potential Clinical Concern in Part 1
Description: Hematology parameters included platelet count, RBC Count, hemoglobin, hematocrit, MCV, MCH, %Reticulocytes, neutrophils, lymphocytes, monocytes, eosinophils, basophils. Clinical chemistry parameters included potassium aspartate aminotransferase(AST)/Serum Glutamic-Oxaloacetic Transaminase (SGOT), total and direct bilirubin, creatinine, sodium alanine, aminotransferase, (ALT)/ Serum Glutamic-Pyruvic, Transaminase (SGPT), total protein, fasting glucose, calcium, alkaline phosphatase and albumin. Urinalysis included specific gravity, potential of hydrogen (pH), glucose, protein, blood and ketones by dipstick and microscopic examination of urine.
Time Frame: Up to 29 days in Part 1
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | 600RC High Fat | 475DC High Fat | 600DC High Fat | 600DC 5%HPMC High Fat | 600RC Fasted | 475DC Fasted | 600DC Fasted | 600DC 5%HPMC Fasted
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

7. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to t (AUC [0-t]) of Danirixin for Part 1
Description: as for outcome 2
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours in Part 1
Population: PK population. Only those participants with data available at specified time points were analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms/milliliter
Arm/Group | 600RC High Fat | 475DC High Fat | 600DC High Fat | 600DC 5%HPMC High Fat | 600RC Fasted | 475DC Fasted | 600DC Fasted | 600DC 5%HPMC Fasted
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 7 | 8 | 8 | 8
Hours*nanograms/milliliter | 5515.9 (24.54) | 5573.6 (17.65) | 5524.7 (22.15) | 5287.0 (28.27) | 11480.1 (28.07) | 10977.2 (30.52) | 10636.5 (32.09) | 11015.8 (28.35)

8. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to 24 Hours Post-dose (AUC [0-24]) of Danirixin for Part 1
Description: as for outcome 2
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours in Part 1
Population: PK population. Only those participants with data available at specified time points were analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms/milliliter
Arm/Group | 600RC High Fat | 475DC High Fat | 600DC High Fat | 600DC 5%HPMC High Fat | 600RC Fasted | 475DC Fasted | 600DC Fasted | 600DC 5%HPMC Fasted
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 7 | 8 | 8 | 8
Hours*nanograms/milliliter | 4919.5 (27.19) | 4952.0 (18.25) | 4984.8 (24.27) | 4705.2 (27.96) | 10744.8 (26.07) | 10419.9 (27.78) | 10029.3 (32.19) | 10319.9 (26.14)

9. Secondary Outcome: Time to Occurrence of Cmax (Tmax) of Danirixin for Part 1
Description: as for outcome 2
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours in Part 1
Population: PK population. Only those participants with data available at specified time points were analyzed
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | 600RC High Fat | 475DC High Fat | 600DC High Fat | 600DC 5%HPMC High Fat | 600RC Fasted | 475DC Fasted | 600DC Fasted | 600DC 5%HPMC Fasted
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 7 | 8 | 8 | 8
Hours | 3.897 (0.9894) | 3.653 (0.5089) | 3.585 (1.2942) | 4.158 (1.3556) | 1.165 (0.3794) | 1.331 (0.7536) | 1.214 (0.2669) | 1.342 (0.3768)

10. Secondary Outcome: Terminal Half-life (t1/2) of Danirixin for Part 1
Description: as for outcome 2
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours in Part 1
Population: PK population. Only those participants with data available at specified time points were analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | 600RC High Fat | 475DC High Fat | 600DC High Fat | 600DC 5%HPMC High Fat | 600RC Fasted | 475DC Fasted | 600DC Fasted | 600DC 5%HPMC Fasted
Number analyzed (Participants) | 5 | 7 | 7 | 6 | 6 | 7 | 8 | 8
Hours | 9.638 (17.60) | 10.904 (19.33) | 8.916 (29.74) | 9.888 (26.18) | 8.298 (36.18) | 9.498 (26.76) | 9.391 (45.40) | 9.107 (29.56)

11. Secondary Outcome: Time to Last Quantifiable Concentration (Tlast) of the Blood Concentration of Danirixin for Part 1
Description: as for outcome 2
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours in Part 1
Population: PK population. Only those participants with data available at specified time points were analyzed
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | 600RC High Fat | 475DC High Fat | 600DC High Fat | 600DC 5%HPMC High Fat | 600RC Fasted | 475DC Fasted | 600DC Fasted | 600DC 5%HPMC Fasted
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 7 | 8 | 8 | 8
Hours | 47.660 (0.2178) | 47.587 (0.2200) | 44.657 (8.3551) | 44.757 (8.3813) | 44.372 (8.9730) | 41.789 (10.9667) | 41.699 (10.9179) | 44.531 (8.3335)

12. Secondary Outcome: Lag Time Before Observation of Drug Concentrations in Sampled Matrix (Tlag) of Danirixin for Part 1
Description: as for outcome 2
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours in Part 1
Population: PK population. Only those participants with data available at specified time points were analyzed
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | 600RC High Fat | 475DC High Fat | 600DC High Fat | 600DC 5%HPMC High Fat | 600RC Fasted | 475DC Fasted | 600DC Fasted | 600DC 5%HPMC Fasted
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 7 | 8 | 8 | 8
Hours | 0.323 (0.3812) | 0.383 (0.5917) | 0.383 (0.5918) | 0.511 (0.6661) | 0.000 (0.000) | 0.065 (0.1830) | 0.000 (0.0000) | 0.000 (0.0000)

13. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to Infinity (AUC [0-inf]) of Danirixin for Part 2
Description: as for outcome 2
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours in Part 2
Population: PK population. Only those participants with data available at specified time points were analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms/milliliter
Groups:
- 475DC-Fasted: Participants received a single dose of DNX 50 mg HBr hemihydrate 475 DC tablet formulation in fasted state
- 475DC-Normal Meal: Participants received DNX 50 mg HBr hemihydrate 475 DC formulation along with normal meal
- 475DC-High Fat: Participants received DNX 50 mg HBr hemihydrate 475 DC formulation along with high fat meal
- 475DC-MONO High Fat: Participants received DNX 50 mg HBr monohydrate 475 DC with 5 percent HPMC formulation along with high fat meal
- 475DC Fasted OMP: Participants received DNX 50 mg HBr hemihydrate 475 DC formulation and OMP under fasted condition
- 475DC Normal Meal OMP: Participants received DNX 50 mg HBr hemihydrate 475 DC formulation and OMP along with normal meal
- 475DC High Fat OMP: Participants received DNX 50 mg HBr hemihydrate 475 DC formulation and OMP along with high fat meal
Arm/Group | 475DC-Fasted | 475DC-Normal Meal | 475DC-High Fat | 475DC-MONO High Fat | 475DC Fasted OMP | 475DC Normal Meal OMP | 475DC High Fat OMP
Number analyzed (Participants) | 12 | 10 | 12 | 11 | 9 | 10 | 7
Hours*nanograms/milliliter | 12426.4 (35.85) | 7761.2 (41.31) | 8136.7 (32.85) | 7356.4 (34.65) | 14615.2 (24.23) | 10185.0 (34.57) | 8782.5 (45.73)

14. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to t (AUC [0-t]) of Danirixin for Part 2
Description: as for outcome 2
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours in Part 2
Population: PK population. Only those participants with data available at specified time points were analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms/milliliter
Arm/Group | 475DC-Fasted | 475DC-Normal Meal | 475DC-High Fat | 475DC-MONO High Fat | 475DC Fasted OMP | 475DC Normal Meal OMP | 475DC High Fat OMP
Number analyzed (Participants) | 12 | 11 | 12 | 12 | 11 | 11 | 11
Hours*nanograms/milliliter | 12026.9 (37.00) | 7484.2 (39.37) | 7757.2 (31.77) | 6986.9 (32.54) | 12903.9 (37.02) | 9023.8 (42.46) | 7885.4 (46.30)

15. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to 24 Hours (AUC [0-24]) of Danirixin for Part 2
Description: as for outcome 2
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours in Part 2
Population: PK population. Only those participants with data available at specified time points were analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms/milliliter
Arm/Group | 475DC-Fasted | 475DC-Normal Meal | 475DC-High Fat | 475DC-MONO High Fat | 475DC Fasted OMP | 475DC Normal Meal OMP | 475DC High Fat OMP
Number analyzed (Participants) | 12 | 11 | 12 | 12 | 10 | 10 | 9
Hours*nanograms/milliliter | 11096.7 (36.64) | 6482.2 (37.93) | 6706.6 (28.49) | 6187.1 (30.41) | 12762.9 (23.58) | 8681.0 (32.68) | 7590.8 (37.96)

16. Secondary Outcome: Maximum Observed Concentration (Cmax) of Danirixin for Part 2
Description: as for outcome 2
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours in Part 2
Population: PK population. Only those participants with data available at specified time points were analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms/milliliter
Arm/Group | 475DC-Fasted | 475DC-Normal Meal | 475DC-High Fat | 475DC-MONO High Fat | 475DC Fasted OMP | 475DC Normal Meal OMP | 475DC High Fat OMP
Number analyzed (Participants) | 12 | 11 | 12 | 12 | 11 | 11 | 11
Nanograms/milliliter | 2317.4 (44.90) | 989.9 (47.91) | 969.9 (37.80) | 1019.8 (38.90) | 2292.5 (43.18) | 1389.7 (43.59) | 1132.5 (35.26)

17. Secondary Outcome: Time to Maximum Observed Concentration (Tmax) of Danirixin for Part 2
Description: as for outcome 2
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours in Part 2
Population: PK population. Only those participants with data available at specified time points were analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | 475DC-Fasted | 475DC-Normal Meal | 475DC-High Fat | 475DC-MONO High Fat | 475DC Fasted OMP | 475DC Normal Meal OMP | 475DC High Fat OMP
Number analyzed (Participants) | 12 | 11 | 12 | 12 | 11 | 11 | 11
Hours | 1.271 (0.3374) | 3.749 (0.6458) | 4.150 (1.5008) | 3.355 (1.3724) | 1.978 (0.8770) | 2.887 (0.7802) | 3.752 (1.7384)

18. Secondary Outcome: Terminal Half-life (t1/2) of Danirixin for Part 2
Description: as for outcome 2
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours in Part 2
Population: PK population. Only those participants with data available at specified time points were analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | 475DC-Fasted | 475DC-Normal Meal | 475DC-High Fat | 475DC-MONO High Fat | 475DC Fasted OMP | 475DC Normal Meal OMP | 475DC High Fat OMP
Number analyzed (Participants) | 12 | 10 | 12 | 11 | 9 | 10 | 7
Hours | 10.647 (26.80) | 11.424 (21.51) | 11.484 (11.21) | 11.652 (20.01) | 11.304 (15.02) | 10.913 (24.37) | 8.975 (33.78)

19. Secondary Outcome: Time to Last Quantifiable Concentration (Tlast) of the Blood Concentration of Danirixin for Part 2
Description: as for outcome 2
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours in Part 2
Population: PK population. Only those participants with data available at specified time points were analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | 475DC-Fasted | 475DC-Normal Meal | 475DC-High Fat | 475DC-MONO High Fat | 475DC Fasted OMP | 475DC Normal Meal OMP | 475DC High Fat OMP
Number analyzed (Participants) | 12 | 11 | 12 | 12 | 11 | 11 | 11
Hours | 45.139 (6.6767) | 47.144 (0.4440) | 47.200 (0.4262) | 46.741 (0.4843) | 45.217 (7.0764) | 45.242 (7.0723) | 40.869 (10.8896)

20. Secondary Outcome: Lag Time Before Observable Concentration (Tlag) of Danirixin for Part 2
Description: as for outcome 2
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 hours in Part 2
Population: PK population. Only those participants with data available at specified time points were analyzed
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | 475DC-Fasted | 475DC-Normal Meal | 475DC-High Fat | 475DC-MONO High Fat | 475DC Fasted OMP | 475DC Normal Meal OMP | 475DC High Fat OMP
Number analyzed (Participants) | 12 | 11 | 12 | 12 | 11 | 11 | 11
Hours | 0.000 (0.0000) | 0.283 (0.3554) | 0.641 (0.4405) | 0.386 (0.4922) | 0.000 (0.0000) | 0.423 (0.3097) | 0.370 (0.6461)

21. Secondary Outcome: Number of Participants With Any Adverse Event (AE) and Serious Adverse Events in Part 2
Description: as for outcome 3
Time Frame: Up to 52 days in Part 2
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | 475DC-Fasted | 475DC-Normal Meal | 475DC-High Fat | 475DC-MONO High Fat | 475DC Fasted OMP | 475DC Normal Meal OMP | 475DC High Fat OMP
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 11 | 11 | 12
Participants
  Any AE | 1 | 1 | 1 | 0 | 0 | 0 | 3
  Any SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Number of Participants With Vital Signs of Potential Clinical Concern in Part 2
Description: as for outcome 4
Time Frame: Up to 52 days in Part 2
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | 475DC-Fasted | 475DC-Normal Meal | 475DC-High Fat | 475DC-MONO High Fat | 475DC Fasted OMP | 475DC Normal Meal OMP | 475DC High Fat OMP
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 11 | 11 | 12
Participants | 2 | 3 | 4 | 4 | 4 | 3 | 4

23. Secondary Outcome: Number of Participants With 12-lead Electrocardiogram (ECG) Values of Potential Clinical Concern in Part 2
Description: Single 12-lead ECGs were obtained using an ECG machine that automatically calculated the heart rate and measured PR, QRS, and QT intervals, and QT interval corrected by Fridericia's formula (QTcF). Number of participants with 12-lead ECG values of potential clinical concern in Part 2 are presented.
Time Frame: Up to 52 days in Part 2
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | 475DC-Fasted | 475DC-Normal Meal | 475DC-High Fat | 475DC-MONO High Fat | 475DC Fasted OMP | 475DC Normal Meal OMP | 475DC High Fat OMP
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 11 | 11 | 12
Participants | 1 | 2 | 1 | 3 | 1 | 2 | 2

24. Secondary Outcome: Number of Participants With Laboratory Values of Potential Clinical Concern in Part 2
Description: Hematology parameters included platelet count, RBC Count, hemoglobin, hematocrit, MCV, MCH, %Reticulocytes, neutrophils, lymphocytes, monocytes, eosinophils, basophils. Clinical chemistry parameters included potassium aspartate, Aminotransferase(AST)/Serum Glutamic-Oxaloacetic Transaminase (SGOT), total and direct, bilirubin, creatinine sodium alanine, Aminotransferase, (ALT)/ Serum Glutamic-Pyruvic, Transaminase (SGPT), total protein, fasting glucose, calcium, alkaline phosphatase and albumin. Urinalysis included specific gravity, potential of hydrogen (pH), glucose, protein, blood and ketones by dipstick and microscopic examination of urine.
Time Frame: Up to 52 days in Part 2
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | 475DC-Fasted | 475DC-Normal Meal | 475DC-High Fat | 475DC-MONO High Fat | 475DC Fasted OMP | 475DC Normal Meal OMP | 475DC High Fat OMP
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 11 | 11 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: On-Treatment serious adverse events (SAEs) and non-serious AEs (nSAEs) were collected from start of study treatment until 81 days
Description: On-Treatment SAEs and nSAEs were reported for mITT Population.
Groups:
- 475DC-Fasted OMP: Participants received DNX 50 mg HBr hemihydrate 475 DC formulation and OMP under fasted condition
- 475DC-Normal Meal OMP: Participants received DNX 50 mg HBr hemihydrate 475 DC formulation and OMP along with normal meal
- 475DC-High Fat OMP: Participants received DNX 50 mg HBr hemihydrate 475 DC formulation and OMP along with high fat meal
Arm/Group | 600RC High Fat | 475DC High Fat | 600DC High Fat | 600DC 5%HPMC High Fat | 600RC Fasted | 475DC Fasted | 600DC Fasted | 600DC 5%HPMC Fasted | 475DC-Fasted | 475DC-Normal Meal | 475DC-High Fat | 475DC-MONO High Fat | 475DC-Fasted OMP | 475DC-Normal Meal OMP | 475DC-High Fat OMP
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/12 | 0/12 | 0/12 | 0/12 | 0/11 | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/12 | 0/12 | 0/12 | 0/12 | 0/11 | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 1/8 | 0/8 | 0/8 | 0/8 | 2/8 | 1/8 | 1/8 | 1/8 | 1/12 | 1/12 | 1/12 | 0/12 | 0/11 | 0/11 | 3/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 600RC High Fat (N=8) | 475DC High Fat (N=8) | 600DC High Fat (N=8) | 600DC 5%HPMC High Fat (N=8) | 600RC Fasted (N=8) | 475DC Fasted (N=8) | 600DC Fasted (N=8) | 600DC 5%HPMC Fasted (N=8) | 475DC-Fasted (N=12) | 475DC-Normal Meal (N=12) | 475DC-High Fat (N=12) | 475DC-MONO High Fat (N=12) | 475DC-Fasted OMP (N=11) | 475DC-Normal Meal OMP (N=11) | 475DC-High Fat OMP (N=12)
Vessel puncture site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-02-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT03457727/Prot_001.pdf
  • Statistical Analysis Plan (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT03457727/SAP_000.pdf